CLINICAL TRIAL: NCT00005783
Title: A Phase I/II Trial of Recombinant-Methionyl Human Stem Cell Factor (SCF) in Adult Patients With Sickling Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000087; 00-DK-0087
Record Dates: First submitted 2000-06-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Hemoglobin SC Disease; Sickle Cell Anemia
Keywords: Fetal Hemoglobin; Hematopoietic Growth Factor; Peripheral Blood CD34 Cells; Vasoocclusive Crisis; Sickle Cell Anemia; Sickle Cell Disease; Sickle Cell Disorder
MeSH Terms: conditions — Hemoglobin SC Disease; Anemia, Sickle Cell; beta-Thalassemia; Vaso-Occlusive Crises | interventions — ancestim

INTERVENTIONS:
Drug: Recombinant-methionyl human stem cell factor

SUMMARY:
Sickle cell anemia is a genetic disorder that results from a single nucleotide substitution in codon 6 of the beta-globin gene which, in the homozygous state, produces an abnormal hemoglobin that is prone to polymer formation when deoxygenated. The polymerized hemoglobin leads to impaired deformability and sickling of red blood cells which subsequently lodge in end-arterioles producing the classic and most prominent feature of the disorder, repeated vasoocclusive crises. Despite knowledge of the precise genetic defect for decades, only recently has there been therapeutic impact based upon this knowledge when a clear benefit from treatment with hydroxyurea, a cell cycle-specific agent administered to induce production of fetal hemoglobin (HbF) by stimulating gamma-globin synthesis, was reported in patients with sickle cell disease (SCD). The reduction in the frequency and severity of vasoocclusive crises seen has been attributed to the increase in HbF levels in responsive patients. While the majority of patients demonstrate a rise in HbF, not all such patients benefit from treatment. Given these results, alternative agents that also stimulate the production of HbF warrant investigation in the treatment of SCD. Recombinant-methionyl human stem cell factor (SCF) is a hematopoietic growth factor with activity on immature hematopoietic progenitor cells. SCF stimulates the production of HbF in vitro and in vivo, and this effect is attainable without the myelosuppression associated with hydroxyurea. In this phase I/II trial, we will administer SCF in a dose escalating fashion to patients with sickling disorders. Parameters to be measured are HbF levels, F cell levels, peripheral blood CD34 levels, frequency, duration, and severity of vasoocclusive crises, and toxicity.

DETAILED DESCRIPTION:
Sickle cell anemia is a genetic disorder that results from a single nucleotide substitution in codon 6 of the beta-globin gene which, in the homozygous state, produces an abnormal hemoglobin that is prone to polymer formation when deoxygenated. The polymerized hemoglobin leads to impaired deformability and sickling of red blood cells which subsequently lodge in end-arterioles producing the classic and most prominent feature of the disorder, repeated vasoocclusive crises. Despite knowledge of the precise genetic defect for decades, only recently has there been therapeutic impact based upon this knowledge when a clear benefit from treatment with hydroxyurea, a cell cycle-specific agent administered to induce production of fetal hemoglobin (HbF) by stimulating gamma-globin synthesis, was reported in patients with sickle cell disease (SCD). The reduction in the frequency and severity of vasoocclusive crises seen has been attributed to the increase in HbF levels in responsive patients. While the majority of patients demonstrate a rise in HbF, not all such patients benefit from treatment. Given these results, alternative agents that also stimulate the production of HbF warrant investigation in the treatment of SCD. Recombinant-methionyl human stem cell factor (SCF) is a hematopoietic growth factor with activity on immature hematopoietic progenitor cells. SCF stimulates the production of HbF in vitro and in vivo, and this effect is attainable without the myelosuppression associated with hydroxyurea. In this phase I/II trial, we will administer SCF in a dose escalating fashion to patients with sickling disorders. Parameters to be measured are HbF levels, F cell levels, peripheral blood CD34 levels, frequency, duration, and severity of vasoocclusive crises, and toxicity.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with Hb SS, Sbeta-thal, SD, or SO-Arab

Age greater than or equal to 18 years.

Patient must have had a previous neurologic event (either symptomatic or found by imaging alone).

More than one painful crises per year for the last 2 years, each requiring hospitalization.

A previous acute chest syndrome.

Evidence of renal damage but with a creatinine clearance of greater than 50 percent of normal.

Red cell alloimmunization.

Bilateral retinopathy.

Osteonecrosis of multiple bones.

Unilateral or bilateral leg ulcers.

Patients who have failed a course of hydroxyurea or who have declined to take hydroxyurea.

Able to give informed consent.

No active sickle cell crises or acute chest syndrome.

No active uncontrolled infection.

No hydroxyurea, erythropoietin, and/or arginine butyrate therapy in the previous month.

No patients receiving hypertransfusion therapy.

No current treatment (or within 2 weeks) with hematopoietic growth factors.

No allergy to E. coli derived products.

No history of seasonal or recurrent asthma within the 5 preceding years.

No asthmatic symptoms (e.g. wheezing) related to a current respiratory tract infection.

No other significant IgE-mediated hypersensitivities (including but not limited to allergic rhinitis, allergic eczema, anaphylactic reactions, congenital or acquired angioedema, and urticaria,). An isolated episode of urticaria occurring within the 5 years is not a contraindication. Patients with drug allergies manifested solely by rash are not excluded.

No concurrent use of beta-adrenergic blocking agents.

No concurrent use of monoamine oxidase inhibitors.

No significant comorbid conditions including uncontrolled hypertension, congestive heart failure(greater NY class II), poorly controlled diabetes mellitus, and significant coronary artery disease with recent myocardial infarction or angioplasty (within the previous 6 months).

No pregnancy, breast feeding, and unwillingness to use contraception.

No concurrent use of other investigational products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2000-03; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States